CLINICAL TRIAL: NCT07132983
Title: A Phase II, Randomized, Double-Blind, Cross-Over Study to Assess the Pharmacokinetics, Pharmacodynamics, and Safety of Single Inhaled Doses of Ensifentrine-Glycopyrrolate Fixed Dose Combination, Ensifentrine, and Glycopyrrolate in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Phase II Study to Assess the Pharmacokinetics, Pharmacodynamics, and Safety of Single Inhaled Doses of Ensifentrine-glycopyrrolate Fixed Dose Combination, Ensifentrine, and Glycopyrrolate in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-CO-210
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; bronchodilator; ensifentrine-glycopyrrolate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A: Ensifentrine plus Glycopyrrolate (Experimental): (fixed-dose combination formulation)
  Subjects will receive a single dose of study medication in each treatment period followed by a 7 to 9-day washout period before receiving the next treatment in the sequence they were assigned to
  Interventions: Drug: Ensifentrine 3 mg; Drug: Glycopyrrolate 42.5 mcg
- Treatment B: Ensifentrine monotherapy (Experimental): (fixed-dose combination formulation)
  Subjects will receive a single dose of study medication in each treatment period followed by a 7 to 9-day washout period before receiving the next treatment in the sequence they were assigned to
  Interventions: Drug: Ensifentrine 3 mg
- Treatment C: Glycopyrrolate monotherapy (Experimental): (fixed-dose combination formulation)
  Subjects will receive a single dose of study medication in each treatment period followed by a 7 to 9-day washout period before receiving the next treatment in the sequence they were assigned to
  Interventions: Drug: Glycopyrrolate 42.5 mcg
- Treatment D: Ensifentrine monotherapy (Experimental): (fixed-dose combination formulation)
  Subjects will receive a single dose of study medication in each treatment period followed by a 7 to 9-day washout period before receiving the next treatment in the sequence they were assigned to
  Interventions: Drug: Ensifentrine 1.5 mg
- Treatment E: Ensifentrine monotherapy (marketed formulation) (Experimental): Subjects will receive a single dose of study medication in each treatment period followed by a 7 to 9-day washout period before receiving the next treatment in the sequence they were assigned to
  Interventions: Drug: Ensifentrine 3 mg (marketed formulation)

INTERVENTIONS:
Drug: Ensifentrine 3 mg — Single dose, administered by oral inhalation using a standard jet nebulizer
  Arms: Treatment A: Ensifentrine plus Glycopyrrolate; Treatment B: Ensifentrine monotherapy
Drug: Glycopyrrolate 42.5 mcg — Single dose, administered by oral inhalation using a standard jet nebulizer
  Arms: Treatment A: Ensifentrine plus Glycopyrrolate; Treatment C: Glycopyrrolate monotherapy
Drug: Ensifentrine 1.5 mg — Single dose, administered by oral inhalation using a standard jet nebulizer
  Arms: Treatment D: Ensifentrine monotherapy
Drug: Ensifentrine 3 mg (marketed formulation) — Single dose, administered by oral inhalation using a standard jet nebulizer
  Arms: Treatment E: Ensifentrine monotherapy (marketed formulation)

SUMMARY:
This study will assess the pharmacokinetics (PK), pharmacodynamics (PD) and safety of ensifentrine and glycopyrrolate fixed dose (FDC) product, the individual components of the FDC (ensifentrine and glycopyrrolate, each in the FDC formulation), ensifentrine 1.5 mg in the FDC formulation and ensifentrine 3 mg in the marketed formulation each administered via a standard jet nebulizer, in adult participants with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Enrolled participants will be expected to participate for approximately 7 weeks: 1 to 2 weeks for screening, 5 single doses of study medication with each dose followed by an approximately 7-day washout period (total of 5 weeks), and 1 week of follow-up. Participants will be randomized to receive all the treatments in different sequences.

The primary objective of the study is to evaluate the pharmacokinetics of the fixed-dose combination of ensifentrine and glycopyrrolate compared to each drug alone and to ensifentrine in a different formulation.

ELIGIBILITY:
Inclusion Criteria:

* Males are eligible to participate if they to use contraception or abstinence, and refrain from donating fresh unwashed semen during the study and for at least 30 days post-study
* Females are eligible to participate if they are not pregnant, breastfeeding and if one of the following conditions apply:

  1. Not a woman of child-bearing potential OR
  2. Agrees to follow the contraceptive guidance and not to donate eggs for the purpose of reproduction from screening throughout the study and for at least 30 days post-study
* Current or former cigarette smokers with a history of cigarette smoking ≥ 10 pack years as of signing the ICF [number of pack years = (number of cigarettes per day / 20) × number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Pipe and/or cigar use cannot be used to calculate pack-year history. Former smokers are defined as those who have stopped smoking for at least 6 months prior to signing the ICF. Smoking cessation programs are permitted during the study
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines with symptoms compatible with COPD
* Post-bronchodilator (4 puffs of albuterol) spirometry during the Screening Period demonstrating both the following:

  1. FEV1/forced vital capacity (FVC) ratio of < 0.70 AND
  2. FEV1 ≥ 40 % and ≤ 80% of predicted normal
* A posterior-anterior chest x-ray (CXR) during the Screening Period or within 12 months prior to signing the ICF showing no clinically significant abnormalities unrelated to COPD. If a CXR within the past 12 months is not available but a computed tomography (CT) scan within the same time period is available, the CT scan may be reviewed in place of a CXR
* Capable of withholding from short-acting bronchodilators for at least 4 hours if using albuterol and for at least 6 hours if using ipratropium prior to pre-dose of blinded study medication spirometry testing
* Anatomical features of peripheral veins that allow the ability to draw sufficient blood volume for all study samples
* Capable of using the study supplied jet nebulizer correctly
* Ability to perform acceptable spirometry in accordance with ATS/ERS guidelines
* Willing and able to attend all study visits and adhere to all study assessments and procedures

Exclusion Criteria:

* Concomitant clinically significant pulmonary disease other than COPD (e.g., asthma, tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, sleep apnea (unless controlled with stable continuous positive airway pressure use), known alpha-1 antitrypsin deficiency, core pulmonale or other non-specific pulmonary disease)
* Within 6 months prior to randomization, a COPD exacerbation requiring hospitalization
* Within 3 months prior to randomization, use of therapies for a COPD exacerbation (e.g., oral, intravenous, or intramuscular glucocorticoids; antibiotics; theophylline; roflumilast)
* History of life-threatening COPD, including Intensive Care Unit admission and/or requiring intubation
* Severe comorbidities including:

  1. Unstable cardiac disease (myocardial infarction within 1 year prior to randomization, unstable angina within 6 months prior to randomization, unstable or life-threatening arrhythmia requiring intervention within 3 months prior to randomization, diagnosis of New York Heart Association (NYHA) class III or IV heart disease)
  2. Any other clinically significant medical conditions including uncontrolled diseases (e.g., endocrine, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric [e.g., untreated significant depression, anxiety, or history of suicidality], or ophthalmic diseases) that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject
* History of or clinically significant on-going bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within 6 months prior to randomization
* History of narrow angle glaucoma
* History of hypersensitivity or intolerance to aerosol medications, albuterol, ensifentrine, glycopyrrolate, any excipients/components of the study medications, anticholinergic agents, or sympathomimetic amines
* History of or current malignancy of any organ system, treated or untreated within the 5 years prior to signing the ICF, except for localized basal or squamous cell carcinoma of the skin
* Other significant psychiatric disease that would likely result in the subject not being able to complete the study, in the opinion of the Investigator
* Findings on physical examination that the Investigator considers to be clinically significant during the Screening Period
* Prior or current use of Ohtuvayre (ensifentrine)
* Previous lung resection or lung reduction surgery within 1-year of randomization
* Patients with a recent history of a COPD exacerbation requiring treatment or hospitalization for an exacerbation are excluded, as are patients requiring supplemental oxygen (defined as oxygen therapy prescribed for the treatment of COPD). As needed oxygen is not exclusionary
* Pulmonary rehabilitation unless such treatment has been stable from 4 weeks prior to signing the ICF and plans to remain stable during the study. Pulmonary rehabilitation programs should not be started or completed during participation in the study
* Major surgery (requiring general anesthesia) in the 6 weeks prior to randomization, lack of full recovery from surgery as of randomization, or planned surgery through the end of the study
* Current or history of drug or alcohol abuse within the 5 years prior to randomization
* Estimated glomerular filtration rate (eGFR) < 30 mL/min as tested during the Screening Period
* Any other abnormal hematology, biochemistry, or viral serology assessed during the Screening Period deemed by the Investigator to be clinically significant
* Alanine aminotransferase (ALT) ≥ 2 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≥ 2 × ULN, alkaline phosphatase and/or total bilirubin > 1.5 × ULN (subjects with Gilbert's syndrome can be included with total bilirubin > 1.5 × ULN as long as direct bilirubin is ≤ 1.5 × ULN)
* Use of an experimental drug within 30 days or 5 half-lives of randomization, whichever is longer, and/or participation in a study treatment-free follow-up phase of a clinical study within 30 days prior to randomization
* Use of an experimental medical device or participation in a follow-up phase of an experimental medical device clinical study within 30 days prior to randomization
* Affiliation with the Investigator site, including an Investigator, Sub-Investigator, study coordinator, study nurse, other employee of participating Investigator or study site or a family member of the aforementioned

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2025-10-06 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Ensifentrine single dose area under the curve from time 0 to time t (AUC0-t) | Day 1 through 48 hours after each dose of study medication
Ensifentrine single dose area under the curve from time 0 extrapolated to infinity (AUC0-inf) | Day 1 through 48 hours after each dose of study medication
Ensifentrine single dose maximum observed concentration (Cmax) | Day 1 through 48 hours after each dose of study medication
Glycopyrronium single dose AUC0-t | Day 1 through 48 hours after each dose of study medication
Glycopyrronium single dose AUC0-inf | Day 1 through 48 hours after each dose of study medication
Glycopyrronium single dose Cmax | Day 1 through 48 hours after each dose of study medication
Change from average baseline in forced expiratory volume over 1 second (FEV1) to FEV1 area under the curve versus time from time 0 to 12 hours (AUC0-12h) | Baseline through 12 hours after each dose of study medication
Change from average baseline FEV1 to average FEV1 area under the curve versus time from time 0 to 4 hours (AUC0-4h) | Baseline through 4 hours after each dose of study medication
Change from average baseline FEV1 to peak FEV1 measured over 4 hours post-dose | Baseline through 4 hours after each dose of study medication
Change from average baseline FEV1 to 12-hour post-dose (evening trough) FEV1 | Baseline through 12 hours after each dose of study medication
Incidence of treatment emergent adverse events (TEAEs) | From first dose through the end of study (approximately 6 weeks)
Change from baseline in QTcF as measured by 12-lead ECG | Baseline and visits 2, 5, 8, 11, and 14
Change from baseline in blood pressure | Baseline through end of study (approximately 6 weeks)
Change from baseline in heart rate | Baseline through end of study (approximately 6 weeks)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Clinical Research of West Florida Inc - Tampa, Tampa, Florida
  - Midwest Chest Consultants PC, Saint Charles, Missouri
  - Velocity Clinical Research - Spartanburg - PPDS, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No